CLINICAL TRIAL: NCT03524027
Title: Posterior Vertebral Column Resection (PVCR) for Correction of Adolescent Thoracolumbar Congenital Kyphoscoliosis (CKS)
Brief Title: Vertebral Column Resection (VCR) in Congenital Kyphoscoliosis (CKS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Muhammad Almessry, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVCR
Record Dates: First submitted 2018-04-26; First posted 2018-05-14 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Congenital Spinal Deformity; Congenital Kyphoscoliosis
Keywords: Vertebral Column Resection; Congenital Spinal Deformity; Congenital Thoracolumbar Kyphoscoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Congenital Thoracolumbar Kyphoscoliosis (Experimental): Correction of Adolescent Thoracolumbar Congenital Kyphoscoliosis (CKS) Spinal Deformity by Posterior Vertebral Column Resection (PVCR) Surgical Technique
  Interventions: Procedure: Posterior Vertebral Column Resection (PVCR)

INTERVENTIONS:
Procedure: Posterior Vertebral Column Resection (PVCR) — Posterior Vertebral Column Resection (PVCR) Surgical Technique for Correction of Adolescent Thoracolumbar Congenital Kyphoscoliosis (CKS) Spinal Deformity
  Other Names: Vertebrectomy; Corpectomy; Spondylectomy; VCR

SUMMARY:
Congenital spinal deformities (CSD) are caused by early embryologic errors in vertebral column formation. Spinal cord malformations are present in approximately one third of patients, even associated cardiac, renal, and genitourinary organ system anomalies in more than half of patients. Functional activity and health-related quality of life (HRQOL) are severely affected in adolescents with neglected severe congenital kyphoscoliosis (CKS) progressive curves in developing countries.

Different strategies are described with two main principles; I- Prophylactic surgeries like hemi-epiphysiodesis or in situ fusions that will cease worsening or allow progressive correction over time, II- Corrective surgeries like reconstructive osteotomies and spinal fusion with or without spinal resection. The perfect show in management of congenital spinal deformities is to pick up the curves at early stages where a prophylactic treatment can be achieved with minimal risk to the spinal cord, but certainly many cases are quite aggressive or come late enough where corrective surgeries and even spinal column resection is the only valid plan.

A posterior-based vertebral column resection (VCR) is considered to be the preferred approach in the treatment of rigid, severe, and complex spinal deformities, however the difficult and lengthy nature of the procedure require assistance from experienced and well trained team. It is relatively safe but challenging technique, that allows for dramatic radiographic correction and clinical improvement. It also carries a complication rate of 10.2% as profound blood loss, iatrogenic neurological deficit and late junctional kyphosis.

DETAILED DESCRIPTION:
Preoperative Details :

Every patient is examined for 1- Shoulder balance 2- Pelvic balance 3- Thoracic hump 4- Neurological examination. Also preoperative whole-spine X-ray anteroposterior and lateral view radiographs in erect position are obtained for accurate preoperative planning. Three-dimensional Multi-Slice Computed Tomography (MSCT) scan is obtained to delineate posterior vertebral column pathoanatomy before surgery. Whole-spine MRI is obtained for declaration of any associated spinal cord malformation.

Operative Details :

Appropriate patient positioning on the operating frame to avoid excessive pressure points in the axilla, allow the abdomen to hang free, and to maintain stability of the trunk during surgery. Standard posterior exposure is performed, and pedicle screws are placed using a free-hand technique as. The exposure at the osteotomy site is extended laterally to resect a portion of the medial ribs to enhance the exposure of the vertebral body to be removed.

Once adequate exposure is achieved, a wide laminectomy is completed from the pedicles of the proximal vertebra to the pedicles of the distal vertebra. Use of tranexamic acid to minimize osseous bleeding during these lengthy surgeries is advisable. At this point, a short rod is placed into the pedicle screws of 1 side to include at least 2 pedicle screws proximally and 2 pedicle screws distally, to provide stability during the osteotomy. Once this rod is secured, the proximal and distal discs are removed and the vertebra to be removed is outlined.

Then, the osteotomy is started from the pedicle on the contralateral side, and extending into the body. The exiting nerve roots are tied and transected at the thoracic levels, gently retracted at the lumbar levels. The removal of vertebral body is proceeded using Kerrison rongeurs and osteotomes as necessary. After adequate removal, another rod is placed to the already osteotomized side, and secured. At this point the rod on the other side can be removed or kept in place, depending on the amount of expected instability.

The resection carried similarly on the contralateral side. The posterior wall of the vertebral body is kept intact until the very end of the osteotomy. After the removal of the vertebral body and discs, using a reverse cutting curette the posterior wall is fractured with anteriorly directed blows and removed using rongeurs. The endplates of the neighboring vertebrae are cleaned off of any remaining cartilage to expose bone surfaces to achieve fusion.

The anterior defect is augmented with morsellized cancellous graft with or without the use of a titanium mesh cage, depending on the width of the void. After the completion of resection, deformity correction is carried out and the posterior instrumentation system is secured using pedicle screws. Application of Wakeup test to detect any on-table neurology. Decortication followed by addition of remaining autograft and allograft to the fusion is performed. Posterior wound closure is performed over a drain.

Postoperative Details :

Follow-up protocol is carried out after 2 weeks, 3 months, 1 year, and 2 years postoperatively with whole-spine X-Ray radiographs in erect position, and after 1 year with Multi-Slice Computed Tomography (MSCT) scan to assess fusion rate.

ELIGIBILITY:
Inclusion Criteria:

* Neglected congenital kyphoscoliotic spinal deformity
* Thoracic and Lumbar curves only
* Age more than 10 years old

Exclusion Criteria:

* Cervical and Sacral deformities
* Revision failed back surgeries

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Change in Scoliosis Research Society (SRS)-24 (arabic version) Health-related quality of life questionnaire | Baseline preoperative, then 3 months, and 1 year postoperative
  The score of questionnaire components is used to assess how patients are doing regarding their function (day to day activities), their pain level (or hopefully improvement in/lack of), how they feel they look, how they feel about themselves, and if they are satisfied as the result of their treatment. Preoperative and postoperative scores are compared.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline preoperative, then 3 months, and 1 year postoperative
  Is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain.
Short Form (SF)-36 Health Survey | Baseline preoperative, then 3 months, and 1 year postoperative
  Is widely validated and popularly used in assessing the subjective quality of life (QOL) of patients and the general public.
Complications Rate | Intraoperative, then Immediate, 2 weeks, 3 months, and 1 year postoperative
  As neurological deficit, vascular injury, deep infection, visual affection, pulmonary embolism, pleural effusion, deep venous thrombosis, implant-related problems, proximal junctional kyphosis, and re-operation for any cause.
American Spinal Injury Association (ASIA) Score | Baseline preoperative, then immediate, and 3 months postoperative
  A score developed by the American Spinal Injury Association for essential minimal elements of neurologic assessment for all patients with a spinal injury.
Local Kyphosis Angle (LKA) | Baseline preoperative, then 2 weeks, and 1 year postoperative
  Assessed on the lateral radiograph by measuring the angle obtained by a line parallel to the inferior endplate of the deformed vertebra and that of the vertebra one level above.
Lumbar Lordosis Angle (LLA) | Baseline preoperative, then 2 weeks, and 1 year postoperative
  Angle measured between L1 and L5 lower end plates.
Thoracic Kyphosis Angle (TKA) | Baseline preoperative, then 2 weeks, and 1 year postoperative
  Angle measured between T1 and T12 lower end plates.
Sagittal Vertical Axis (SVA) to C7 Plumb Line (C7PL) | Baseline preoperative, then 2 weeks, and 1 year postoperative
  To quantify global alignment. It is defined as the sagittal offset of a plumb line dropped from the C7 vertebral body from the posterosuperior corner of the sacral plate.
Scoliosis Angle (Cobb's Angle) | Baseline preoperative, then 2 weeks, and 1 year postoperative
  To measure and quantify the magnitude of spinal deformities, especially in the case of scoliosis. The Cobb angle measurement is the "gold standard" of scoliosis evaluation endorsed by Scoliosis Research Society. It is used as the standard measurement to quantify and track the progression of scoliosis.
Shoulder Balance (Clavicle Angle) | Baseline preoperative, then 2 weeks, and 1 year postoperative
  It is the angle that is subtended between a horizontal reference line - clavicle horizontal reference line (CHRL), which is drawn perpendicular to the lateral edge of the radiograph and touches the most cephalad portion of the elevated clavicle and a line which touches the most cephalad aspect of both the right and left clavicles - clavicle reference line (CRL). By convention, angles subtended with the left shoulder up are positive and angles subtended with the right shoulder up are negative (consistent with directionality of the T1 tilt angle).
Central Sacral Vertical Line (CSVL) to C7 Plumb Line (C7PL) | Baseline preoperative, then 2 weeks, and 1 year postoperative
  Coronal decompensation is measured as the horizontal distance between a plumb line dropped downward from the center of the C7 (C7PL) vertebral body and the central sacral vertical line (CSVL), which is a line drawn vertically through the center of the sacrum.
Body Height (BH) | Baseline preoperative, then 2 weeks, and 1 year postoperative
  The height is measured using a measuring tape with patient standing without shoes.
T1-S1 Trunk Height (TH) | Baseline preoperative, then 2 weeks, and 1 year postoperative
  The T1-S1 height of the spine and the T1-S1 length of the spine are measured and compared.
Leg Length Discrepancy (LLD) | Baseline preoperative, then 1 year postoperative
  Radiographic measurement of difference between the lengths of the legs. Full-length standing anteroposterior radiograph compared with scanogram.
CT-based Classification for assessment of biological graft fusion | 1 year postoperative
  A new assessment method of bony union using high-speed spiral CT imaging is proposed which reflects the gradually increasing biological stability of the construct. Grade I (complete fusion) implies cortical union of the allograft and central trabecular continuity. Grade II (partial fusion) implies cortical union of the structural allograft with partial trabecular incorporation. Grade III (unipolar pseudarthrosis) denotes superior or inferior cortical non-union of the central allograft with partial trabecular discontinuity centrally and Grade IV (bipolar pseudarthrosis) suggests both superior and inferior cortical non-union with a complete lack of central trabecular continuity.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed El-Meshtawy, Study Chair — Assiut University; Belal Elnady, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aydogan M, Ozturk C, Tezer M, Mirzanli C, Karatoprak O, Hamzaoglu A. Posterior vertebrectomy in kyphosis, scoliosis and kyphoscoliosis due to hemivertebra. J Pediatr Orthop B. 2008 Jan;17(1):33-7. doi: 10.1097/01.bpb.0000218031.75557.f0. PMID 18043375
- [Background] Lenke LG, O'Leary PT, Bridwell KH, Sides BA, Koester LA, Blanke KM. Posterior vertebral column resection for severe pediatric deformity: minimum two-year follow-up of thirty-five consecutive patients. Spine (Phila Pa 1976). 2009 Sep 15;34(20):2213-21. doi: 10.1097/BRS.0b013e3181b53cba. PMID 19752708
- [Background] Ayvaz M, Akalan N, Yazici M, Alanay A, Acaroglu RE. Is it necessary to operate all split cord malformations before corrective surgery for patients with congenital spinal deformities? Spine (Phila Pa 1976). 2009 Oct 15;34(22):2413-8. doi: 10.1097/BRS.0b013e3181b9c61b. PMID 19829255
- [Background] Ruf M, Jensen R, Letko L, Harms J. Hemivertebra resection and osteotomies in congenital spine deformity. Spine (Phila Pa 1976). 2009 Aug 1;34(17):1791-9. doi: 10.1097/BRS.0b013e3181ab6290. PMID 19644330
- [Background] Hedequist D, Emans J. Congenital scoliosis. J Am Acad Orthop Surg. 2004 Jul-Aug;12(4):266-75. doi: 10.5435/00124635-200407000-00007. PMID 15473678
- [Background] Soliman HAG. Health-related Quality of Life of Adolescents With Severe Untreated Congenital Kyphosis and Kyphoscoliosis in a Developing Country. Spine (Phila Pa 1976). 2018 Aug;43(16):E942-E948. doi: 10.1097/BRS.0000000000002598. PMID 29462064
- [Background] Wang Y, Lenke LG. Vertebral column decancellation for the management of sharp angular spinal deformity. Eur Spine J. 2011 Oct;20(10):1703-10. doi: 10.1007/s00586-011-1771-0. Epub 2011 Mar 19. PMID 21424339
- [Background] Lenke LG, Shaffrey CI, Carreon LY, Cheung KMC, Dahl BT, Fehlings MG, Ames CP, Boachie-Adjei O, Dekutoski MB, Kebaish KM, Lewis SJ, Matsuyama Y, Mehdian H, Pellise F, Qiu Y, Schwab FJ; AO Spine International and SRS Scoli-RISK-1 Study Group. Lower Extremity Motor Function Following Complex Adult Spinal Deformity Surgery: Two-Year Follow-up in the Scoli-RISK-1 Prospective, Multicenter, International Study. J Bone Joint Surg Am. 2018 Apr 18;100(8):656-665. doi: 10.2106/JBJS.17.00575. PMID 29664852
- [Background] Lenke LG, Sides BA, Koester LA, Hensley M, Blanke KM. Vertebral column resection for the treatment of severe spinal deformity. Clin Orthop Relat Res. 2010 Mar;468(3):687-99. doi: 10.1007/s11999-009-1037-x. Epub 2009 Sep 1. PMID 19727995
- [Background] Lenke LG, Newton PO, Sucato DJ, Shufflebarger HL, Emans JB, Sponseller PD, Shah SA, Sides BA, Blanke KM. Complications after 147 consecutive vertebral column resections for severe pediatric spinal deformity: a multicenter analysis. Spine (Phila Pa 1976). 2013 Jan 15;38(2):119-32. doi: 10.1097/BRS.0b013e318269fab1. PMID 22825478